CLINICAL TRIAL: NCT06053606
Title: The Impact of Cryoablation Using Expandable (POLARxFIT) vs. Standard Size (POLARx) Balloon on Autonomic Control of the Heart
Brief Title: The Impact of Expandable Cryoballoon on Autonomic Control of the Heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Piotr Niewinski, MD, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POLARxFIT and GPs
Record Dates: First submitted 2023-09-17; First posted 2023-09-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation; ganglionated plexus; autonomic modulation; cryoablation; cryoballoon; expandable balloon
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- expandable cryoballoon (Experimental): POLARxFIT
  Interventions: Device: cryoablation of atrial fibrillation using expandable balloon (28 / 31 mm)
- standard cryoballoon (Experimental): POLARx
  Interventions: Device: cryoablation of atrial fibrillation using only 28 mm size balloon

INTERVENTIONS:
Device: cryoablation of atrial fibrillation using only 28 mm size balloon — all applications in all PVs are done with 28 mm balloon
  Arms: standard cryoballoon
Device: cryoablation of atrial fibrillation using expandable balloon (28 / 31 mm) — first applications in LSPV and RSPV are done with 31 mm balloon
  Arms: expandable cryoballoon

SUMMARY:
Approximately 40% of patients following cryoballoon ablation show signs of parasympathetic denervation. The presence of such effect is related to better outcomes in terms of clinical efficacy (freedom from atrial fibrillation). It could be hypothesized that larger sized balloon (POLARxFIT system) because of more antral position within the left atrium (and hence smaller distance from ganglionated plexi) might enhance this beneficial modulation of the autonomic system of the heart. This study intends to compare the effects of cryoablation employing expandable balloon (POLARxFIT) vs. standard balloon (POLARx) on autonomic system of the heart.

ELIGIBILITY:
Inclusion Criteria:

* primary PVI
* paroxysmal atrial fibrillation
* sinus rhythm at the admission
* participant meets clinical criteria for PVI

Exclusion Criteria:

* LA diameter <38 mm or >50 mm
* LVEF <40%
* intrinsic sinus node disease
* advanced atrioventricular block (PR interval >300 ms, II or III degree AV block)
* previous cardioneuroablation procedure
* pregnancy
* contraindications to anticoagulation treatment
* any other clinical contraindications to PVI
* known atropine intolerance

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
difference in the rate of persistent parasympathetic modulation | 3 months
  defined as decrease in RR interval of >20%

SECONDARY OUTCOMES:
difference in time to first AF episode | 12 months
  days
difference in left atrial dwell time | periprocedural
  minutes
difference in radiation dose | periprocedural
  mGy
difference in contrast volume | periprocedural
  mililiters

OTHER OUTCOMES:
occurence of persistent phrenic nerve palsy | periprocedural
  event rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Niewinski, MD, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Institute of Heart Diseases, Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Time Frame: after study completion
Access Criteria: upon reasonable request